CLINICAL TRIAL: NCT01288976
Title: ACCESS-Europe A Two-Phase Observational Study of the MitraClip® System in Europe
Acronym: ACCESS-EU
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: EU-0901
Record Dates: First submitted 2011-01-25; First posted 2011-02-03 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Mitral Valve (MV) Regurgitation
Keywords: Mitral Valve; Mitral Regurgitation; MitraClip; Mitral Valve Surgery; Mitral Valve Insufficiency or Mitral Regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux; Mitral Valve Insufficiency | interventions — Practice Management, Medical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MitraClip Therapy: Patients treated with the MitraClip System.
  Interventions: Device: MitraClip
- Medical Management: Patients with MR managed non-surgically based on standard hospital clinical practice.
  Interventions: Drug: Medical Management
- Mitral Valve Surgery: Patients with MR managed surgically (repair or replacement) based on standard hospital clinical practice.
  Interventions: Procedure: Mitral Valve Surgery

INTERVENTIONS:
Device: MitraClip — The MitraClip System includes a MitraClip device, a Steerable Guide Catheter, and a MitraClip Delivery System that enables placement of the MitraClip device on the mitral valve leaflets
  Groups: MitraClip Therapy
Drug: Medical Management — The Non-Surgical Medically Managed Heart Failure (HF) Group consists of patients with mitral regurgitation (MR) in whom the MR is managed non-surgically based on standard hospital clinical practice. Patients with MR who receive a pacemaker, Implantable Cardiac Defibrillator (ICD) and/or Cardiac Resynchronization Therapy (CRT) treatments may be included
  Groups: Medical Management
Procedure: Mitral Valve Surgery — The Mitral Valve Surgery Group consists of patients with MR in whom the MR is managed surgically (repair or replacement) based on standard hospital clinical practice. Patients with concurrent coronary artery bypass grafting (CABG) or aortic/tricuspid valve or and other cardiac procedure except atrial fibrillation surgery are excluded.
  Groups: Mitral Valve Surgery

SUMMARY:
The MitraClip System enables the European physicians an alternative therapeutic option for patients with mitral regurgitation (MR). Therapeutic alternatives are open-heart cardiac surgery, and palliative medical therapy with or without device therapy. The study will observe the outcomes of patients treated with the MitraClip System throughout 12-months as compared to the outcomes of patients treated by alternative therapies.

DETAILED DESCRIPTION:
PHASE I:

The primary objective of ACCESS-EU Phase I is to gain information in the European Union Countries regarding the use of the MitraClip System with respect to health economics and clinical care.

PHASE II: (HAS BEEN CLOSED BY SPONSOR) The primary objective of ACCESS-EU Phase II is to gather additional clinical data, specifically Echocardiography Core Laboratory measurements of MR severity and left ventricular volumes and diameters, and other echocardiographic measures, on patients undergoing the MitraClip procedure in the European Union Countries,

Clinical data collected from both study phases, is expected to contribute to decision making with regards to MitraClip therapy selection in patients with MR: (a) by establishing the value of the MitraClip therapy in the continuum of care; and (b) by providing practical information that will allow physicians to make therapeutic decisions, assist hospitals to make purchasing decisions, and assist insurers in making coverage decisions.

Study Design:

ACCESS-Europe is a two-phase prospective, observational, multicenter post-approval study of the MitraClip System for the treatment of mitral regurgitation (MR) in the European Union Countries. Patients will be evaluated per standard practice at baseline, discharge, 6-Months and 12-Months.

Phase I of the study consists of patients who receive the MitraClip system for the treatment of MR and two concurrent comparator groups of (a) medically managed heart failure patients with MR and (b) patients who have undergone mitral valve surgery for MR. The two comparator groups will be followed and evaluated primarily from a health economic perspective.

ACCESS EU Study Phase II will consist of only patients who receive the MitraClip System, with the objective to collect additional clinical data, specifically Echocardiography Core Laboratory evaluation of MR severity and other echocardiographic measures.

Enrollment of patients in each study phase is as follows:

ACCESS-EU PHASE I:

* A minimum of 300 MitraClip Therapy group patients,
* A minimum of 100 patients in the Mitral Valve Surgery comparator group
* As many patients as possible in the Medical Therapy comparator group

First Patient Enrollment Projection: Q1, 2009 Last Patient Enrollment Projection: Enrollment in the Mitral Valve Surgery and Medically Therapy groups ceased on December 31, 2010. Enrollment in the MitraClip group will cease when Phase II of the study is initiated at each site.

ACCESS-EU PHASE II:

A minimum of 300 MitraClip therapy subjects will be enrolled in Phase II.

First Patient Enrollment Projection: Q2, 2011 Last Patient Enrollment Projection: Enrollment will cease when the Sponsor has determined that an adequate number of patients have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Per the current approved labeling for the Conformity European (CE) Marked MitraClip System.

Exclusion Criteria:

* Per the current approved labeling for the CE Marked MitraClip System.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Mitral Regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 721 (Actual)
Dates: Start 2008-10; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, PhD, Study Director — Abbott Vascular Structural Heart (Evalve Inc); Wolfgang Schillinger, MD, Principal Investigator — Universitatsmedizin Gottingen; Francesco Maisano, MD, Principal Investigator — Fondazion Ctr San Raffaele Del Monte Tabor Istituto
Locations (1):
- Universitatsmedizin Gottingen, Göttingen, Germany

REFERENCES:
- [Background] Rogers JH, Yeo KK, Carroll JD, Cleveland J, Reece TB, Gillinov AM, Rodriguez L, Whitlow P, Woo YJ, Herrmann HC, Young JN. Late surgical mitral valve repair after percutaneous repair with the MitraClip system. J Card Surg. 2009 Nov-Dec;24(6):677-81. doi: 10.1111/j.1540-8191.2009.00901.x. Epub 2009 Jul 24. PMID 19682161
- [Background] Feldman T, Kar S, Rinaldi M, Fail P, Hermiller J, Smalling R, Whitlow PL, Gray W, Low R, Herrmann HC, Lim S, Foster E, Glower D; EVEREST Investigators. Percutaneous mitral repair with the MitraClip system: safety and midterm durability in the initial EVEREST (Endovascular Valve Edge-to-Edge REpair Study) cohort. J Am Coll Cardiol. 2009 Aug 18;54(8):686-94. doi: 10.1016/j.jacc.2009.03.077. PMID 19679246
- [Background] Herrmann HC, Kar S, Siegel R, Fail P, Loghin C, Lim S, Hahn R, Rogers JH, Bommer WJ, Wang A, Berke A, Lerakis S, Kramer P, Wong SC, Foster E, Glower D, Feldman T; EVEREST Investigators. Effect of percutaneous mitral repair with the MitraClip device on mitral valve area and gradient. EuroIntervention. 2009 Jan;4(4):437-42. doi: 10.4244/eijv4i4a76. PMID 19284064
- [Background] Luk A, Butany J, Ahn E, Fann JI, St Goar F, Thornton T, McDermott L, Madayag C, Komtebedde J. Mitral repair with the Evalve MitraClip device: histopathologic findings in the porcine model. Cardiovasc Pathol. 2009 Sep-Oct;18(5):279-85. doi: 10.1016/j.carpath.2008.07.001. Epub 2008 Aug 13. PMID 18703359
- [Background] Silvestry FE, Rodriguez LL, Herrmann HC, Rohatgi S, Weiss SJ, Stewart WJ, Homma S, Goyal N, Pulerwitz T, Zunamon A, Hamilton A, Merlino J, Martin R, Krabill K, Block PC, Whitlow P, Tuzcu EM, Kapadia S, Gray WA, Reisman M, Wasserman H, Schwartz A, Foster E, Feldman T, Wiegers SE. Echocardiographic guidance and assessment of percutaneous repair for mitral regurgitation with the Evalve MitraClip: lessons learned from EVEREST I. J Am Soc Echocardiogr. 2007 Oct;20(10):1131-40. doi: 10.1016/j.echo.2007.02.003. Epub 2007 Jun 13. PMID 17570634
- [Background] Borgia F, Di Mario C, Franzen O. Adenosine-induced asystole to facilitate MitraClip placement in a patient with adverse mitral valve morphology. Heart. 2011 May;97(10):864. doi: 10.1136/hrt.2010.208132. Epub 2010 Oct 29. No abstract available. PMID 21036802
- [Background] Tamburino C, Imme S, Barbanti M, Mule M, Pistritto AM, Aruta P, Cammalleri V, Scarabelli M, Mangiafico S, Scandura S, Ussia GP. Reduction of mitral valve regurgitation with Mitraclip(R) percutaneous system. Minerva Cardioangiol. 2010 Oct;58(5):589-98. PMID 20948505
- [Background] Ciobanu A, Bennett S, Azam M, Clark A, Vinereanu D. Incremental value of three-dimensional transoesophageal echocardiography for guiding double percutaneous MitraClip (R) implantation in a 'no option' patient. Eur J Echocardiogr. 2011 Feb;12(2):E11. doi: 10.1093/ejechocard/jeq118. Epub 2010 Sep 27. PMID 20876188
- [Background] Lim DS, Kunjummen BJ, Smalling R. Mitral valve repair with the MitraClip device after prior surgical mitral annuloplasty. Catheter Cardiovasc Interv. 2010 Sep 1;76(3):455-9. doi: 10.1002/ccd.22547. PMID 20839359
- [Background] Kalarus Z, Kukulski T, Lekston A, Streb W, Sikora J, Nadziakiewicz P, Gasior M, Polonski L, Zembala M. [Methodology and safety of transvascular reduction of severe ischaemic mitral insufficiency with MitraClip in high-surgical-risk patients - first three cases in Poland]. Kardiol Pol. 2010 Jun;68(6):729-35. Polish. PMID 20806217
- [Background] Geidel S, Ostermeyer J, Lass M, Schmoeckel M. Complex surgical valve repair after failed percutaneous mitral intervention using the MitraClip device. Ann Thorac Surg. 2010 Jul;90(1):277-9. doi: 10.1016/j.athoracsur.2009.12.048. PMID 20609795
- [Background] Mauri L, Garg P, Massaro JM, Foster E, Glower D, Mehoudar P, Powell F, Komtebedde J, McDermott E, Feldman T. The EVEREST II Trial: design and rationale for a randomized study of the evalve mitraclip system compared with mitral valve surgery for mitral regurgitation. Am Heart J. 2010 Jul;160(1):23-9. doi: 10.1016/j.ahj.2010.04.009. PMID 20598968
- [Background] Jonsson A, Settergren M. MitraClip catheter-based mitral valve repair system. Expert Rev Med Devices. 2010 Jul;7(4):439-47. doi: 10.1586/erd.10.23. PMID 20583881
- [Background] Ussia GP, Barbanti M, Tamburino C. Feasibility of percutaneous transcatheter mitral valve repair with the MitraClip system using conscious sedation. Catheter Cardiovasc Interv. 2010 Jun 1;75(7):1137-40. doi: 10.1002/ccd.22415. PMID 20336809
- [Background] Tamburino C, Ussia GP, Maisano F, Capodanno D, La Canna G, Scandura S, Colombo A, Giacomini A, Michev I, Mangiafico S, Cammalleri V, Barbanti M, Alfieri O. Percutaneous mitral valve repair with the MitraClip system: acute results from a real world setting. Eur Heart J. 2010 Jun;31(11):1382-9. doi: 10.1093/eurheartj/ehq051. Epub 2010 Mar 18. PMID 20299349
- [Background] Franzen O, Baldus S, Rudolph V, Meyer S, Knap M, Koschyk D, Treede H, Barmeyer A, Schofer J, Costard-Jackle A, Schluter M, Reichenspurner H, Meinertz T. Acute outcomes of MitraClip therapy for mitral regurgitation in high-surgical-risk patients: emphasis on adverse valve morphology and severe left ventricular dysfunction. Eur Heart J. 2010 Jun;31(11):1373-81. doi: 10.1093/eurheartj/ehq050. Epub 2010 Mar 10. PMID 20219746
- [Background] Argenziano M, Skipper E, Heimansohn D, Letsou GV, Woo YJ, Kron I, Alexander J, Cleveland J, Kong B, Davidson M, Vassiliades T, Krieger K, Sako E, Tibi P, Galloway A, Foster E, Feldman T, Glower D; EVEREST Investigators. Surgical revision after percutaneous mitral repair with the MitraClip device. Ann Thorac Surg. 2010 Jan;89(1):72-80; discussion p 80. doi: 10.1016/j.athoracsur.2009.08.063. PMID 20103209
- [Result] Maisano F, Franzen O, Baldus S, Schafer U, Hausleiter J, Butter C, Ussia GP, Sievert H, Richardt G, Widder JD, Moccetti T, Schillinger W. Percutaneous mitral valve interventions in the real world: early and 1-year results from the ACCESS-EU, a prospective, multicenter, nonrandomized post-approval study of the MitraClip therapy in Europe. J Am Coll Cardiol. 2013 Sep 17;62(12):1052-1061. doi: 10.1016/j.jacc.2013.02.094. Epub 2013 Jun 7. PMID 23747789
- [Result] Ussia GP, Cammalleri V, Scandura S, Imme S, Pistritto AM, Ministeri M, Chiaranda M, Caggegi A, Barbanti M, Aruta P, Tamburino C. Update on percutaneous mitral valve therapy: clinical results and real life experience. Minerva Cardioangiol. 2012 Feb;60(1):57-70. PMID 22322574
- [Result] Maisano F, Godino C, Giacomini A, Denti P, Buzzatti N, Arendar I, Colombo A, Alfieri O, La Canna G. Patient selection for MitraClip therapy impaired left ventricular systolic function. Minerva Cardioangiol. 2011 Oct;59(5):455-71. PMID 21983306
- [Derived] Blazek S, Lurz P, Mangner N, Fuernau G, Seeburger J, Luecke C, Gutberlet M, Ender J, Desch S, Eitel I, Schuler G, Thiele H. Incidence, characteristics and functional implications of cerebral embolic lesions after the MitraClip procedure. EuroIntervention. 2015 Feb;10(10):1195-203. doi: 10.4244/EIJY14M05_10. PMID 24831647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The ACCESS-EU Phase I Study began enrolling patients in October 2, 2008 and completed enrollment on April 13, 2011. There were 567 patients enrolled at 14 investigational sites in Europe. The last follow-up visit occurred on June 15, 2012 and the last monitoring visit occurred August 9, 2012.
Groups:
- Medical Management: Patients with MR managed nonsurgically based on standard hospital clinical practice. Medical Management: The NonSurgical Medically Managed Heart Failure (HF) Group consists of patients with mitral regurgitation (MR) in whom the MR is managed nonsurgically based on standard hospital clinical practice. Patients with MR who receive a pacemaker, Implantable Cardiac Defibrillator (ICD) and/or Cardiac Resynchronization Therapy (CRT) treatments may be included.
- Mitral Valve Surgery: Patients with MR managed surgically (repair or replacement) based on standard hospital clinical practice. Mitral Valve Surgery: The Mitral Valve Surgery Group consists of patients with MR in whom the MR is managed surgically (repair or replacement) based on standard hospital clinical practice. Patients with concurrent coronary artery bypass grafting (CABG) or aortic/tricuspid valve or and other cardiac procedure except atrial fibrillation surgery are excluded.
Period: Overall Study
Arm/Group | MitraClip Therapy | Medical Management | Mitral Valve Surgery
Started | 567 | 49 | 105
Completed | 389 | 22 | 85
Not Completed | 178 | 27 | 20
Not completed — Withdrawal by Subject | 58 | 12 | 9
Not completed — Death | 98 | 6 | 4
Not completed — Data unavailable | 22 | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MitraClip Therapy | Medical Management | Mitral Valve Surgery | Total
Number analyzed (Participants) | 567 | 49 | 105 | 721
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (9.6) | 70.7 (12.6) | 60.0 (15.2) | 68.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 23 | 46 | 274
  Male | 362 | 26 | 59 | 447
Region of Enrollment [Number; unit: participants]
  Europe | 567 | 49 | 105 | 721

OUTCOME MEASURES:

1. Primary Outcome: MR Severity
Description: MR Severity: Site-assessed mitral regurgitation severity using echocardiography. MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 1+ to 2+ is mild-to-moderate, 2+ to 3+ is moderate to moderate-to-Severe, 3+ is moderate-to-severe, 3+ to 4+ is moderate-to-severe to severe, 4+ is severe.
  MR severity was not consistently captured for patients in the Medical Management and Mitral Valve Surgery groups. The Medical Therapy & Mitral Valve Surgery comparator groups were followed & studied primarily from a health economic perspective. Availability of clinical outcomes at followup is limited & has not been validated. Clinical outcomes for the comparator groups will not be reported.
Time Frame: At baseline
Population: MR severity was not consistently captured for patients in the Medical Management and Mitral Valve Surgery groups. MR severity will not be reported for these comparator arms. A total of 240 patients excluded from analysis population due to death:98, withdrew consent:58, lost to follow-up:22 and missed mitral regurgitation evaluation:62 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 327
percentage of participants
  0:None | 0.0
  1+:Mild | 0.0
  1+ to 2+: Mild-to-Moderate | 0.0
  2+:Moderate | 3.1
  2+ to 3+: Moderate to Moderate-to-Severe | 9.2
  3+:Moderate-to-Severe | 35.8
  3+ to 4+: Moderate-to-Severe to Severe | 21.7
  4+:Severe | 30.3

2. Primary Outcome: MR Severity
Description: MR Severity: Site-assessed mitral regurgitation severity using echocardiography. MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 1+ to 2+ is mild-to-moderate, 2+ to 3+ is moderate to moderate-to-Severe, 3+ is moderate-to-severe, 3+ to 4+ is moderate-to-severe to severe, 4+ is severe.
  MR severity was not consistently captured for patients in the Medical Management and Mitral Valve Surgery groups. The Medical Therapy & Mitral Valve Surgery comparator groups were followed & studied primarily from a health economic perspective. Availability of clinical outcomes at follow-up is limited & has not been validated. Clinical outcomes for the comparator groups will not be reported.
Time Frame: At 12 months
Population: MR severity was not consistently captured for patients in the Medical Management and Mitral Valve Surgery groups. MR severity will not be reported for these comparator arms. A total of 240 patients excluded from analysis population due to death:98, withdrew consent:58, lost to follow-up:22 and missed mitral regurgitation evaluation:62 at 12 months.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 327
percentage of participants
  0:None | 2.8
  1+:Mild | 27.8
  1+ to 2+: Mild-to-Moderate | 15.0
  2+: Moderate | 33.3
  2+ to 3+: Moderate to Moderate-to-Severe | 9.8
  3+: Moderate-to-Severe | 6.7
  3+ to 4+: Moderate-to-Severe to Severe | 1.5
  4+: Severe | 3.1

3. Secondary Outcome: Procedure Time
Description: Procedure Time is defined as the time of start of the transseptal procedure to the time the Steerable Guide Catheter is removed.
Time Frame: Day 0 (On the day of procedure)
Population: Procedure time is reported only for patients who underwent the MitraClip procedure. This outcome measure does not apply to the Medical Management or the Mitral Valve Surgery groups.
  Procedure Time was not recorded for 196 of 567 patients.Therefore, the data is available for 371 patients.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 371
Minutes | 116.9 (68.1)

4. Secondary Outcome: Contrast Volume
Time Frame: Day 0 (On the day of procedure)
Population: Contrast volume is reported only for patients who underwent the MitraClip procedure. This outcome measure does not apply to the Medical Management or the Mitral Valve Surgery groups.
  Contrast volume was not recorded for 9 of 567 patients. Therefore, Contrast volume is available for 558 subjects.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 558
milliliter | 17.0 (39.7)

5. Secondary Outcome: Fluoroscopy Duration
Time Frame: Day 0 (On the day of procedure)
Population: Fluoroscopy duration is reported only for patients who underwent the MitraClip procedure. This outcome measure does not apply to the Medical Management or the Mitral Valve Surgery groups
  Fluoroscopy duration was not recorded for 99 of 567 patients. Therefore, Fluoroscopy duration is available for 468 patients
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 468
Minutes | 29.1 (19.8)

6. Secondary Outcome: Number of MitraClip Devices Implanted
Description: Physicians had the option of deploying more than 1 MitraClip device if a single device did not provide satisfactory MR reduction, and if the mitral valve area was large enough to allow multiple MitraClip devices to be placed without causing mitral stenosis.
Time Frame: Day 0 (On the day of procedure)
Population: Number of MitraClip Devices Implanted is reported only for patients who underwent the MitraClip procedure.The Medical Therapy&Mitral Valve Surgery comparator groups were followed&studied primarily from a health economic perspective. Availability of clinical outcomes for the comparator groups is limited, thus it has not been validated and reported.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 567
percentage of participants
  0 MitraClip Devices | 0.4
  1 MitraClip Devices | 60.1
  2 MitraClip Devices | 36.7
  3 MitraClip Devices | 2.6
  4 MitraClip Devices | 0.2

7. Secondary Outcome: ICU and Hospital Stay
Description: ICU and hospital stay is defined as the mean duration of time that patients spent in the ICU (Intensive Care Unit)/ CCU (Cardiac Care Unit)/ PACU (Post-Anesthesia Care Unit) following the MitraClip procedure. This secondary outcome measure does not apply to the Medical Management or the Mitral Valve Surgery groups.
Time Frame: From the day of procedure throughout 12 months of study period
Population: ICU and Hospital Stay is reported only for patients who underwent the MitraClip procedure.The Medical Therapy&Mitral Valve Surgery comparator groups were followed&studied primarily from a health economic perspective. Availability of clinical outcomes for the comparator groups is limited, thus it has not been validated and reported.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 567
Days
  Post-procedure ICU/CCU/PACU Duration (n=567) | 2.5 (6.5)
  Post-procedure hospital stay (n=564) | 7.7 (8.2)

8. Secondary Outcome: Discharge Status and Facility
Time Frame: At discharge, an average of 7.7 days following the MitraClip procedure
Population: Discharge Status and Facility is reported only for patients who underwent the MitraClip procedure. This secondary outcome measure does not apply to the Medical Management or the Mitral Valve Surgery groups.Discharge Status and Facility outcomes data is available for 563 patients.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 563
percentage of participants
  Death | 2.0
  Home without home health care | 79.2
  Home with home health care | 0.4
  Skilled nursing facility/ Hospital | 17.1
  Nursing home | 1.4

9. Secondary Outcome: Discharge MR Severity
Time Frame: At discharge, an average of 7.7 days following the MitraClip procedure
Population: MR severity was not consistently captured for patients in the Medical Management and Mitral Valve Surgery groups.MR severity will not be reported for these comparator arms.
  A total of 521 MitraClip patients analyzed.Missing data is due to death(n=11),patient withdrawal(n=13),data unavailable(n=3),discharge echocardiogram not done/missing(n=19).
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 521
percentage of participants
  0:None | 4.4
  1+:Mild | 46.4
  1+ to 2+: Mild-to-Moderate | 14.0
  2+:Moderate | 26.3
  2+ to 3+:Moderate to Moderate-to-Severe | 4.4
  3+:Moderate-to-Severe | 3.1
  3+ to 4+:Moderate-to-Severe to Severe | 1.0
  4+:Severe | 0.4

10. Secondary Outcome: Kaplan-Meier Freedom From All-Cause Mortality
Time Frame: At 0 day
Population: Kaplan-Meier freedom from all-cause mortality is not reported for the Medical Management or the Mitral Valve Surgery groups comparator groups. Since they were followed&studied primarily from a health economic perspective. Availability of clinical outcomes for the comparator groups is limited, thus it has not been validated and reported.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 567
percentage of participants | 100.0

11. Secondary Outcome: Kaplan-Meier Freedom From All-Cause Mortality
Time Frame: At 30 days
Population: Kaplan-Meier freedom from all-cause mortality is not reported for the Medical Management or the Mitral Valve Surgery groups comparator groups. Since they were followed & studied primarily from a health economic perspective. Availability of clinical outcomes for the comparator groups is limited, thus it has not been validated and reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 567
percentage of participants | 96.6 [94.7 to 97.8]

12. Secondary Outcome: Kaplan-Meier Freedom From All-Cause Mortality
Time Frame: At 6 months
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 567
percentage of participants | 88.2 [85.1 to 90.6]

13. Secondary Outcome: Kaplan-Meier Freedom From All-Cause Mortality
Time Frame: At 12 months
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 567
percentage of participants | 81.8 [78.1 to 84.8]

14. Secondary Outcome: Device Embolization and Single Leaflet Device Attachment
Description: Device embolization is defined as bilateral Clip detachment resulting in Clip embolization. Reasons for Clip embolization include leaflet tearing, Clip unlocking, Clip fracture or inadequate Clip placement (i.e., malposition). Not included are any fractures or other failures of the Clip that do not result in Clip detachment from both leaflets.
  Single leaflet device attachment (SLDA) is defined as the loss of insertion of a single leaflet from the MitraClip device with ongoing insertion of the opposing leaflet. SLDAs are reported on ACCESS-EU adverse event log and MitraClip procedure electronic case report forms, and may also be reported by Abbott Vascular personnel per EU Vigilance requirements.
Time Frame: Through 12 months
Population: Device Embolization and Single Leaflet Device Attachment are reported only for patients who underwent the MitraClip procedure. This outcome measure does not apply to the Medical Management or the Mitral Valve Surgery groups.
Measure: Number; unit: participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 567
participants
  Device embolization | 0
  SLDA | 27

15. Secondary Outcome: 1-Day Post-Procedure Safety Outcomes
Description: This outcome measure does not apply to the Medical Management or the Mitral Valve Surgery groups. Because the Medical Therapy&Mitral Valve Surgery comparator groups were followed&studied primarily from a health economic perspective.Availability of clinical outcomes at follow-up is limited & has not been validated. Clinical outcomes for the comparator groups will not be reported.
Time Frame: On day 1 post procedure
Population: 1-Day Post-Procedure Safety Outcomes are reported only for patients who underwent the MitraClip procedure. This outcome measure does not apply to the Medical Management or the Mitral Valve Surgery groups
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 567
percentage of participants
  Death | 0
  Stroke | 0
  Myocardial Infarction | 0.2
  Respiratory Failure | 0
  Need for Resuscitation | 1.1
  Cardiac Tamponade | 0.9
  Mitral Valve Surgery | 0.7

16. Secondary Outcome: Need for Mitral Valve Surgery
Description: This end point is assessed on subjects who underwent mitral valve surgery within 12 months post-MitraClip procedure.
Time Frame: Through 12 months
Population: This outcome measure is reported only for the MitraClip device group. The need for mitral valve surgery was not captured in the Medical Management or the Mitral Valve Surgery groups.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 567
percentage of participants | 6.3

17. Secondary Outcome: NYHA Functional Class
Description: New York Heart Association (NYHA) Functional Classification.
  Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest.Ordinary physical activity results in fatigue, palpitation, dyspnea or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.Less than ordinary physical activity causes fatigue, palpitation dyspnea or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest.If any physical activity is undertaken,discomfort is increased.
Time Frame: At baseline
Population: NYHA Functional Class was not consistently captured for patients in the Medical Management&Mitral Valve Surgery groups.NYHA Functional Class will not be reported for these comparator arms.A total of 567 MitraClip patients,343 analyzed due to death:98,withdrew consent:58,lost to follow-up:22,patients had missing NYHA Functional Class assessment:46 .
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 343
percentage of participants
  NYHA I | 1.7
  NYHA II | 16
  NYHA III | 72.3
  NYHA IV | 9.9

18. Secondary Outcome: NYHA Functional Class
Description: Defined as assessment of NYHA functional class status at follow-up compared to baseline NYHA functional class status.
  Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity.Patients are comfortable at rest.Ordinary physical activity results in fatigue, palpitation, dyspnea/anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity.They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea/anginal pain Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken,discomfort is increased.
Time Frame: At 12 month
Population: NYHA Functional Class was not consistently captured for patients in the Medical Management&Mitral Valve Surgery groups.NYHA Functional Class will not be reported for these comparator arms.Of total 567 MitraClip patients,343 analyzed due to death:98,withdrew consent:58,lost to follow-up:22,patients had missing NYHA Functional Class assessment:46 .
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 343
percentage of participants
  NYHA I | 25.1
  NYHA II | 46.4
  NYHA III | 26.8
  NYHA IV | 1.7

19. Secondary Outcome: The Change in 6 Minute Walk Test Distance From Baseline to 12 Months
Description: The 6 minute walk distance test will be used to measure the patient's exercise capacity. The change in 6 minute walk test distance is calculated as the difference between the distance walked at 12 months and the distanced walked at baseline.
Time Frame: Baseline and 12 months
Population: The 6-minute walk test was not consistently captured for patients in the Medical Management&Mitral Valve Surgery groups.Thus it will not be reported for these comparator arms.Of the 567 MitraClip device patients,216 analyzed due to death:98,withdrew consent:58,lost to follow-up:22&173 patients did not perform the 6-minute walk test.
  .
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 216
meters
  Baseline | 274.7 (118.7)
  12 months | 334.2 (127.9)
  Improvement from Baseline to 12 Months | 59.5 (112.4)

20. Secondary Outcome: Change in Minnesota Living With Heart Failure (MLWHF) Quality of Life Score From Baseline to 12 Months
Description: The Minnesota Living with Heart Failure Questionnaire(MLHFQ) is comprised of 21 questions.The response for each question ranges from 0(no affect on the patient's living) to 5(affected the patient's life very much during the past month).The total score for the 21 items can range from 0-105.A lower&higher MLHFQ score indicates less effect of heart failure&the worse impact of heart failure on a patient's QOL,respectively.Although the MLHFQ incorporates relevant aspects of the key dimensions of QOL (physical and emotional),the questionnaire was not designed to measure any particular dimension separately.The total score should be taken as the best measure of how heart failure and treatments impact QOL.
  The total score is the sum of a)the physical dimension,measured using 8 questions (possible subscale score range 0-40) b)the emotional dimension,measured using 5 questions(possible subscale score from 0-25)&c) other factors,measured using 8 questions (possible subscale score from 0-40).
Time Frame: 12 months
Population: The MLWHF Questionnaire was not consistently administered to patients in the Medical Management&Mitral Valve Surgery groups.Thus MLWHF will not be reported for these comparator arms.Of the 567 MitraClip device patients,264 analyzed due to death:98,withdrew consent:58,lost to follow-up:22&125 patients did not complete MLWHF Questionnaire.
Measure: Mean (Standard Deviation); unit: Quality of Life Score
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 264
Quality of Life Score
  Baseline | 41.6 (18.9)
  12 months | 28.1 (20.1)
  Difference (12 Months - Baseline) | -13.5 (20.5)

21. Secondary Outcome: Six Minute Walk Test Distance (6MWT)
Description: The 6-minute walk distance test will be used to measure the patient's exercise capacity.
Time Frame: Baseline
Population: The 6-minute walk test was not consistently captured for patients in the Medical Management&Mitral Valve Surgery groups.Thus it will not be reported for these comparator arms.Of the 567 MitraClip device patients,216 analyzed due to death:98,withdrew consent:58,lost to follow-up:22&173 patients did not perform the 6-minute walk test at baseline.
  .
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 216
meters | 274.7 (118.7)

22. Secondary Outcome: Six Minute Walk Test Distance (6MWT)
Description: The 6-minute walk distance test will be used to measure the patient's exercise capacity.
Time Frame: 12 months
Population: The 6-MWT was not consistently captured for patients in the Medical Management&Mitral Valve Surgery groups.Thus it will not be reported for these comparator arms.Of the 567 MitraClip device patients,216 analyzed due to death:98,withdrew consent:58,lost to follow-up:22&173 patients did not perform the 6-minute walk test at the12 month visit.
  .
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitraClip Therapy
Number analyzed (Participants) | 216
meters | 334.2 (127.9)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | MitraClip Therapy | Medical Management | Mitral Valve Surgery
All-Cause Mortality (participants affected / at risk) | 13/567 | 1/49 | 2/105
Serious Adverse Events (participants affected / at risk) | 371/567 | 21/49 | 58/105
Other Adverse Events (participants affected / at risk) | 367/567 | 20/49 | 56/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip Therapy (N=567) | Medical Management (N=49) | Mitral Valve Surgery (N=105)
Atrial Septal Defect (ASD) (Cardiac disorders) | 15 (16) | 0 (0) | 0 (0)
Arteriovenous (AV) fistula Fistula (Cardiac disorders) | 6 (6) | 0 (0) | 0 (0)
Atrioventricular block (AV block) (Cardiac disorders) | 6 (6) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 57 (69) | 1 (1) | 8 (8)
Angina (Cardiac disorders) | 13 (14) | 0 (0) | 1 (1)
Aortic Valve (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Arrhythmia, Other (Cardiac disorders) | 26 (26) | 4 (5) | 5 (5)
Arrhythmias (Cardiac disorders) | 13 (15) | 0 (0) | 5 (5)
Ascites (Gastrointestinal disorders) | 9 (12) | 0 (0) | 0 (0)
Atrial arrhythmias (Cardiac disorders) | 45 (55) | 5 (6) | 20 (25)
Bacteremia/Septicemea (Infections and infestations) | 12 (12) | 0 (0) | 2 (2)
Bleeding complications (Vascular disorders) | 26 (26) | 0 (0) | 1 (1)
Blood pressure complications (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Bone and Joint Injuries (Musculoskeletal and connective tissue disorders) | 7 (9) | 0 (0) | 0 (0)
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 76 (94) | 1 (1) | 0 (0)
Bronchial and Lung disorders (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) | 0 (0)
Bruise/Contusion/Ecchymosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (CAD) (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 7 (8) | 1 (1) | 2 (2)
Cardiac: Other (Cardiac disorders) | 31 (32) | 1 (1) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 5 (6) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 14 (14) | 2 (2) | 0 (0)
Cerebro-vascular : Other (Nervous system disorders) | 10 (10) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 7 (7) | 0 (0) | 3 (3)
Coagulopathology (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (non-productive) (General disorders) | 3 (3) | 0 (0) | 0 (0)
Death (General disorders) | 13 (13) | 1 (1) | 2 (2)
Device complications (Injury, poisoning and procedural complications) | 18 (19) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Edema (Vascular disorders) | 45 (49) | 0 (0) | 2 (2)
Endocarditis (Cardiac disorders) | 4 (4) | 0 (0) | 2 (2)
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0) | 0 (0)
Epistaxis (General disorders) | 3 (3) | 0 (0) | 0 (0)
Esophageal injury (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders (Eye disorders) | 6 (6) | 0 (0) | 0 (0)
Fever (General disorders) | 12 (12) | 1 (1) | 0 (0)
Gastrointestinal (GI) hemorrhage (Gastrointestinal disorders) | 12 (18) | 0 (0) | 0 (0)
Gastrointestinal (GI) Infection (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Gastrointestinal (GI) : Other (Gastrointestinal disorders) | 22 (22) | 1 (1) | 5 (5)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal motility (Gastrointestinal disorders) | 13 (13) | 0 (0) | 0 (0)
Generalized pain (General disorders) | 12 (14) | 0 (0) | 0 (0)
Generalized weakness/fatigue (General disorders) | 18 (21) | 2 (2) | 1 (1)
Heart Failure (Cardiac disorders) | 98 (138) | 3 (5) | 1 (3)
Hematologic Miscellaneous (Blood and lymphatic system disorders) | 40 (43) | 3 (3) | 2 (2)
Hematoma: Other (Vascular disorders) | 24 (26) | 0 (0) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoptysis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 10 (10) | 1 (1) | 2 (2)
Hypervolemia (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 14 (14) | 1 (1) | 4 (4)
Hypovolemia (Vascular disorders) | 5 (5) | 0 (0) | 0 (0)
Infections (Infections and infestations) | 16 (16) | 0 (0) | 5 (5)
Mental disorders (Psychiatric disorders) | 17 (17) | 0 (0) | 1 (1)
Metabolic/Endocrine disorders (Metabolism and nutrition disorders) | 42 (47) | 5 (5) | 2 (3)
Miscellaneous (General disorders) | 8 (8) | 0 (0) | 0 (0)
Mitral Valve (Cardiac disorders) | 34 (34) | 1 (1) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal other (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 1 (1) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 5 (5) | 0 (0) | 2 (2)
Nausea (General disorders) | 10 (10) | 0 (0) | 0 (0)
Miscellaneous:other (General disorders) | 55 (63) | 4 (4) | 6 (6)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 33 (37) | 2 (2) | 4 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 3 (3) | 2 (2)
Pseudoaneurysm (Vascular disorders) | 5 (5) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 47 (53) | 2 (2) | 7 (7)
Renal: Other (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal/Urinary Infection (Renal and urinary disorders) | 27 (30) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Retroperitoneal hematoma (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Skin infections (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Stroke (ischemic or hemorrhagic) (Vascular disorders) | 6 (6) | 0 (0) | 0 (0)
Syncope and dizziness (General disorders) | 21 (22) | 2 (3) | 1 (2)
Transient ischemic attack (TIA) (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 7 (7) | 0 (0) | 1 (1)
Tricuspid Valve (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Urinary Miscellaneous (Renal and urinary disorders) | 13 (15) | 0 (0) | 0 (0)
Vascular : other (Vascular disorders) | 22 (24) | 0 (0) | 2 (2)
Ventricular arrhythmias (Cardiac disorders) | 24 (25) | 2 (2) | 0 (0)
Lower respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip Therapy (N=567) | Medical Management (N=49) | Mitral Valve Surgery (N=105)
Atrial Septal Defect (ASD) (Cardiac disorders) | 15 (16) | 0 (0) | 0 (0)
Arteriovenous (AV) fistula Fistula (Cardiac disorders) | 6 (6) | 0 (0) | 0 (0)
Atrioventricular block (AV block) (Cardiac disorders) | 6 (6) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 57 (69) | 1 (1) | 8 (8)
Angina (Cardiac disorders) | 13 (14) | 0 (0) | 1 (1)
Aortic Valve (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Arrhythmia, Other (Cardiac disorders) | 26 (26) | 4 (5) | 5 (5)
Arrhythmias (Cardiac disorders) | 13 (15) | 0 (0) | 5 (5)
Ascites (Gastrointestinal disorders) | 9 (12) | 0 (0) | 0 (0)
Atrial arrhythmias (Cardiac disorders) | 45 (55) | 5 (6) | 20 (25)
Bacteremia/Septicemea (Infections and infestations) | 12 (12) | 0 (0) | 2 (2)
Bleeding complications (Vascular disorders) | 26 (26) | 0 (0) | 1 (1)
Blood pressure complications (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Bone and Joint Injuries (Musculoskeletal and connective tissue disorders) | 7 (9) | 0 (0) | 0 (0)
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 76 (94) | 1 (1) | 0 (0)
Bronchial and Lung disorders (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) | 0 (0)
Bruise/Contusion/Ecchymosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (CAD) (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 7 (8) | 1 (1) | 2 (2)
Cardiac: Other (Cardiac disorders) | 31 (32) | 1 (1) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 5 (6) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 14 (14) | 2 (2) | 0 (0)
Cerebrovascular : Other (Nervous system disorders) | 10 (10) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 7 (7) | 0 (0) | 3 (3)
Coagulopathology (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (non-productive) (General disorders) | 3 (3) | 0 (0) | 0 (0)
Device complications (Injury, poisoning and procedural complications) | 18 (19) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Edema (Vascular disorders) | 45 (49) | 0 (0) | 2 (2)
Endocarditis (Cardiac disorders) | 4 (4) | 0 (0) | 2 (2)
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0) | 0 (0)
Epistaxis (General disorders) | 3 (3) | 0 (0) | 0 (0)
Esophageal injury (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders (Eye disorders) | 6 (6) | 0 (0) | 0 (0)
Fever (General disorders) | 12 (12) | 1 (1) | 0 (0)
Gastrointestinal (GI) hemorrhage (Gastrointestinal disorders) | 12 (18) | 0 (0) | 0 (0)
Gastrointestinal (GI) Infection (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Gastrointestinal (GI) : Other (Gastrointestinal disorders) | 22 (22) | 1 (1) | 5 (5)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal motility (Gastrointestinal disorders) | 13 (13) | 0 (0) | 0 (0)
Generalized pain (General disorders) | 12 (14) | 0 (0) | 0 (0)
Generalized weakness/fatigue (General disorders) | 18 (21) | 2 (2) | 1 (1)
Heart Failure (Cardiac disorders) | 98 (138) | 3 (5) | 1 (3)
Hematologic Miscellaneous (Blood and lymphatic system disorders) | 40 (43) | 3 (3) | 2 (2)
Hematoma: Other (Vascular disorders) | 24 (26) | 0 (0) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoptysis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 10 (10) | 1 (1) | 2 (2)
Hypervolemia (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 14 (14) | 1 (1) | 4 (4)
Hypovolemia (Vascular disorders) | 5 (5) | 0 (0) | 0 (0)
Infections (Infections and infestations) | 16 (16) | 0 (0) | 5 (5)
Mental disorders (Psychiatric disorders) | 17 (17) | 0 (0) | 1 (1)
Metabolic/Endocrine disorders (Metabolism and nutrition disorders) | 42 (47) | 5 (5) | 2 (3)
Miscellaneous (General disorders) | 8 (8) | 0 (0) | 0 (0)
Mitral Valve (Cardiac disorders) | 34 (34) | 1 (1) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal other (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 1 (1) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 5 (5) | 0 (0) | 2 (2)
Nausea (General disorders) | 10 (10) | 0 (0) | 0 (0)
Miscellaneous : other (General disorders) | 55 (63) | 4 (4) | 6 (6)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 33 (37) | 2 (2) | 4 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 3 (3) | 2 (2)
Pseudoaneurysm (Vascular disorders) | 5 (5) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 47 (53) | 2 (2) | 7 (7)
Renal: Other (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal/Urinary Infection (Renal and urinary disorders) | 27 (30) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Retroperitoneal hematoma (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Skin infections (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Stroke (ischemic or hemorrhagic) (Vascular disorders) | 6 (6) | 0 (0) | 0 (0)
Syncope and dizziness (General disorders) | 21 (22) | 2 (3) | 1 (2)
Transient ischemic attack (TIA) (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 7 (7) | 0 (0) | 1 (1)
Tricuspid Valve (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Urinary Miscellaneous (Renal and urinary disorders) | 13 (15) | 0 (0) | 0 (0)
Vascular : other† (Vascular disorders) | 22 (24) | 0 (0) | 2 (2)
Ventricular arrhythmias (Cardiac disorders) | 24 (25) | 2 (2) | 0 (0)
Lower respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days